CLINICAL TRIAL: NCT06598046
Title: A Single-arm, Prospective Phase Ⅱ Clinical Study of Utidelone Combined with Capecitabine in the Treatment of Active Brain Metastasis of Triple-negative Advanced Breast Cancer.
Brief Title: A Single-arm, Prospective Phase Ⅱ Clinical Study of Utidelone Combined with Capecitabine in the Treatment of Active Brain Metastasis of TNBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Min Yan, MD, Principal Investigator, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-MBC15-BM06
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One arm involving utidelone and capecitabine (Experimental): Combination use of utidelone and capecitabine Utidelone 30 mg/m2 d1-5(single-day dose allowed ± 10% fluctuation) , once every three weeks; capecitabine: 1000 mg/m2, twice daily, orally after meal (one in the morning and one in the evening, with an interval of about 12 hours, equivalent to a daily dose of 2000 mg/m2) ; The drug was administered consecutively on days 1-14, with a 21-day cycle.
  Interventions: Drug: Utidelone and capecitabine

INTERVENTIONS:
Drug: Utidelone and capecitabine — Utidelone: intravenous capecitabine: oral

SUMMARY:
This study aims to explore the efficacy and safety of the combination therapy of utidelone and capecitabine in the treatment of brain metastases from triple-negative advanced breast cancer, and to search for systemic treatment for brain metastases from triple-negative advanced breast cancer cases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Invasive breast cancer confirmed by histological or cytological examination, accompanied by metastatic disease; Patients with metastatic diseases not confirmed by pathology or cytology should obtain clear evidence of metastasis through physical examination or radiological research;
3. Based on the pathological report of recent biopsy or other pathological specimens (confirmed by the laboratory of the participating research center), the histology and/or cytology are confirmed as triple negative breast cancer. The specific requirements include: a) the definition of negative human epidermal growth factor receptor 2(HER2): the immunohistochemistry (IHC) is 0 or 1+; If IHC was 2+, it was confirmed negative by fluorescence in situ hybridization (FISH). B) Negative estrogen and progesterone receptors means that IHC examination shows ER < 10% and or PR < 10%, and the researcher evaluates that patients cannot benefit from endocrine therapy.
4. Newly diagnosed brain metastases or brain metastases that have progressed after local treatment: patients with brain metastases who met all the criteria of this scheme before starting from September 1, 2023 and did not meet all the exclusion criteria can also be included;
5. Patients must have measurable central nervous system diseases, defined as at least one brain parenchymal lesion, which can be accurately measured in at least one dimension through local radiological examination; And there is no central nervous system symptom or symptom controllable, so radiotherapy is not needed urgently.
6. Patients who have previously received at least one taxane and/or one anthracycline antibiotic (as a treatment history of neoadjuvant therapy, adjuvant therapy or metastatic therapy or both);
7. Allow (new) adjuvant therapy to have recurrence and metastasis after stopping using Utterone and/or Capecitabine for more than one year, or stop taking drugs for non-progressive reasons in the rescue stage;
8. The physical status score (ECOGPS) of the eastern cancer cooperative group is 0-2, and the life expectancy is more than 12 weeks;
9. Normal organ and bone marrow function; Blood routine examination was basically normal within one week before joining the group (based on the normal laboratory of each research center): neutrophil count (ANC) ≥ 1.5× 109/L; Hemoglobin (HB) ≥ 90g/L; Platelet count (PLT) ≥ 75× 109/L; Liver and kidney function tests were basically normal within one week before enrollment (based on the normal values of laboratories in each research center): total bilirubin (TBIL)≤1.5× upper limit of normal value (ULN); Alanine aminotransferase (SGPT/ALT)≤2.5×ULN (patients with liver metastasis ≤ 5 XULN); Aspartate aminotransferase (SGOT/AST)≤2.5× upper limit of normal value (ULN); Creatinine clearance rate (Ccr)≥60ml/min.
10. Neuropathy should be < grade 2 within 4 weeks before enrollment (version 5.0 of ncictcae);
11. No major organ dysfunction and no heart disease;
12. Women and male patients with reproductive potential must agree to use appropriate contraceptive measures before the start of the study and during the study participation.

Exclusion Criteria:

1. Patients with extensive meningeal metastasis and brain metastasis who are ineffective in dehydration treatment with hormones or in urgent need of radiotherapy;
2. Invasive breast cancer confirmed by histological or cytological examination, accompanied by metastatic disease; Patients with metastatic diseases not confirmed by pathology or cytology should obtain clear evidence of metastasis through physical examination or radiological research;
3. Received chemotherapy, major surgery, targeted therapy or immunotherapy within 2 weeks before joining the group (the interval between targeted therapy and immunotherapy is at least 2 weeks or at least 5 half-lives, whichever is shorter); Received endocrine therapy within 1 week before joining the group; He had received nitrosourea or mitomycin chemotherapy within 6 weeks before joining the group;
4. Receive unlisted clinical trial drugs within 4 weeks before entering the group;
5. Previous history of grade 3 or 4 allergic reactions related to Utterone or Capecitabine;
6. inability to swallow, chronic diarrhea and intestinal obstruction, there are many factors that affect the taking and absorption of drugs;
7. Known contraindications for gadolinium MRI contrast agents, such as pacemakers, shrapnel or ocular foreign bodies;
8. Suffering from other malignant tumors in the past 3 years, excluding cured cervical carcinoma in situ, basal cell carcinoma of skin, squamous cell carcinoma of skin or early thyroid carcinoma;
9. Seizures occurred more than 2 times within 4 weeks before joining the group;
10. Poor control of hypertension; Or have a history of hypertensive crisis or hypertensive encephalopathy;
11. Have a history of bleeding in the central nervous system of grade 3 or above within 12 months;
12. Suffering from serious or uncontrollable diseases, including but not limited to: 1) active virus infection, such as HIV and HBV active phase (HbsAg positive and HBV-DNA≥103, hepatitis C antibody positive); 2) Suffering from severe cardiovascular disease in the past: uncontrollable hypertension; Myocardial infarction, unstable arrhythmia, congestive heart failure, pericarditis, myocarditis, etc. According to NYHA criteria, patients with grade Ⅲ ~ Ⅳ cardiac insufficiency, or those with left ventricular ejection fraction (LVEF) less than 50% indicated by echocardiography; 12. Suffering from serious or uncontrollable diseases, including but not limited to: 1) active virus infection, such as HIV and HBV active phase (HbsAg positive and HBV-DNA≥103, hepatitis C antibody positive); 2) Suffering from severe cardiovascular disease in the past: uncontrollable hypertension; Myocardial infarction, unstable arrhythmia, congestive heart failure, pericarditis, myocarditis, etc. According to NYHA criteria, patients with grade Ⅲ ~ Ⅳ cardiac insufficiency, or those with left ventricular ejection fraction (LVEF) less than 50% indicated by echocardiography;
13. Have a history of hemoptysis within 6 months before joining the group; Or evidence of bleeding tendency or obvious coagulation dysfunction in the last month;
14. Currently receiving full-dose warfarin or equivalent drugs, or taking aspirin (325mg/ day) within 10 days; 15.28 days or in the course of the study, it is expected that major surgery, open biopsy or major trauma are needed;

16. Those who have a history of abdominal fistula or gastrointestinal perforation in the first 6 months; There are unhealed wounds, active ulcers or untreated fractures; Pregnant or lactating women; 17. Those who have a history of psychotropic substance abuse and cannot quit or patients with mental disorders; 18. According to the judgment of the researcher, there are other patients with accompanying diseases that seriously endanger the safety of patients or affect the completion of the study; 19. Those who are known to have allergic history to the drug components of this scheme; Have a history of immunodeficiency, including HIV positive, HCV or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation; 20. The history of live attenuated vaccine inoculation within 28 days before the first study or the person who is expected to be vaccinated with live attenuated vaccine in the study; 21. Any situation that the researcher thinks is not suitable for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
CNS-ORR（RANO Standard） | From the date of enrollment to the date of first documented progression or death from any cause, whichever comes first，assessed up to 48 months.
  CNS-ORR（RANO Standard）

SECONDARY OUTCOMES:
CNS-ORR (RECIST1.1 standard) | From the date of enrollment to the date of first documented progression or death from any cause, whichever comes first，assessed up to 48 months.
  CNS-ORR (RECIST1.1 standard)
CNS-PFS assessed by the investigator | From the date of enrollment to the date of first documented progression or death from any cause, whichever comes first，assessed up to 48 months.
  CNS-PFS assessed by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Breast Cancer Center, The Affiliated Cancer Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No